CLINICAL TRIAL: NCT05076916
Title: Development and Evaluation of the Effectiveness of the Web-based Education Programme Among Cancer Patients Undergoing Treatment of Systemic Chemotherapy: A Randomised Controlled Trial
Brief Title: The Effectiveness of the Web-based Education Programme Among Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Hicran Bektas, PhD, Professor, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2520
Record Dates: First submitted 2021-09-29; First posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Web-based Intervention; Cancer
Keywords: Cancer; Nursing; Self Efficacy; Symptom Management; Quality of Life; Web-Based Education
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: The effect of the web-based education program on patient outcomes was analyzed by dividing the participants into groups through randomization. All patients with cancer who met the sampling criteria were assigned to the intervention and control groups through block randomization (1:1). The web-based education program was introduced to the patients with cancer in the intervention group during face-to-face interviews. They were asked to examine the program for at least two hours a week for three months. During the follow-up period, the patients in the intervention group were called twice a week and reminded to use the education program. The researchers get in contact with the patients online via the website. During the follow-up period, the patients contact the research team by calling or writing messages via the website 24/7.
  The control group received routine patient education and routine hospital follow-ups given by Oncology Education Nurses during the three-month follow-up period.
Who Masked: Participant
Masking Description: For assigning each patient to a group, the subjects were assigned to the groups according to the randomization list created. Two independent researchers conducted the assignment of the participants on the intervention and control groups and the evaluation of the outcome measurement data. Since the researchers conducted the interventions, they were not be blinded. However, the participants were blinded because they did not know the hypotheses of the study and which group they were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The web-based education program was introduced to the patients with cancer in the intervention group during face-to-face interviews. They were asked to examine the program for at least two hours a week for three months. During the follow-up period, the patients in the intervention group were called twice a week and reminded to use the education program. The researchers get in contact with the patients online via the website. During the follow-up period, the patients contact the research team by calling or writing messages via the website 24/7. An e-mail account was created by the research team using the email system of the university, and it was shared with the patients. The clinical researchers of the team answered the patients' questions via this e-mail account. In the third month, after the follow-up stage of the study was completed, the post-tests were administered to the patients in the intervention group who came to the hospital for follow-up or treatment.
  Interventions: Behavioral: The effectiveness of the web-based education programme among cancer patients
- Control group (No Intervention): The control group received routine patient education and routine hospital follow-ups given by Oncology Education Nurses during the three-month follow-up period. In the third month, after the follow-up stage of the study was completed, the post-tests were administered to the patients in the control group who came to the hospital for follow-up or treatment.

INTERVENTIONS:
Behavioral: The effectiveness of the web-based education programme among cancer patients — The web-based education program was introduced to the patients with cancer in the intervention group during face-to-face interviews. They were asked to examine the program for at least two hours a week for three months. During the follow-up period, the patients in the intervention group were called twice a week and reminded to use the education program. The researchers get in contact with the patients online via the website. The patients contact the research team by calling or writing messages via the website 24/7. An e-mail account was created by the research team using the email system of the university, and it was shared with the patients. The clinical researchers of the team answered the patients' questions via this e-mail account.
  Arms: Intervention group

SUMMARY:
This study aims to develop a web-based education program among cancer patients undergoing treatment of systemic chemotherapy and to evaluate the effect of the program on symptom control, quality of life, self-efficacy, and depression. Evaluating the effect of the web-based education programme among cancer patients will be useful in planning appropriate remote nursing interventions to increase the symptom control and quality of life of patients.

A web-based education program was prepared in line with patient needs, evidence-based guidelines, and expert opinions and tested with 10 cancer patients. A single-blind, randomised controlled study design was applied. Pre-tests were applied to 60 cancer patients undergoing systemic chemotherapy, and the patients (intervention:30, control: 30) were randomized. The intervention group used the web-based education program for three months, and they were allowed to communicate with the researchers 24/7 via the website. The effectiveness of the web-based education program at baseline and after 12 weeks evaluated.

DETAILED DESCRIPTION:
Cancer is a life-threatening disease with negative physical, psychological, and socioeconomic effects. Patients with cancer receive outpatient chemotherapy and must manage the most important symptoms of chemotherapy at home without the support of a healthcare professional. Patients with cancer and their families need to be supported not only in the hospital but also in the home environment. Patients want to receive information about strategies for coping with symptoms or problems that they encounter frequently after treatment. It has been reported that the rate of use and effectiveness of web-based programs planned by determining the needs of patients with cancer will be higher. Although experimental studies examining the effect of health education and counseling conducted on the web are limited, no web-based education program created by evaluating the needs of patients with cancer has been found. Our study was conducted to determine the needs of patients with cancer for a web-based education program and to design a program to meet the needs.

The primary aim of the study is to develop a web-based education program for patients with cancer receiving systemic treatment and to test the validity of this program. The secondary aim is to evaluate the effect of this web-based education program on symptom control, quality of life, self-efficacy, and depression in patients with cancer undergoing systemic chemotherapy.

In the first stage of the study, the needs of patients for web-based education were determined using a descriptive design, and in the second stage, the effectiveness of the web-based education program was evaluated using a randomized controlled trial design, with the participants being single-blinded. A randomized controlled trial based on the Consolidated Standard of Reporting Trials - CONSORT 2010 - guidelines was performed.

In the first stage of the study, 30 patients with cancer were interviewed to determine their expectations regarding their needs for web-based education. In the second stage of the study, the sample size was calculated on the G*POWER software package based on an 85% power and a 5% confidence interval. The study was conducted with patients with cancer (n=60), including 30 in the intervention and 30 in the control groups. The study consisted of patients who were over the age of 18, received at least two cycles of systemic chemotherapy, had no verbal communication disorder, were literate, had Internet access and use the Internet. Data of both stages of the study were collected between May 7, 2014, and February 17, 2016.

The effect of the web-based education program on patient outcomes was analyzed by dividing the participants into groups through randomization. All patients with cancer who met the sampling criteria were assigned to the intervention and control groups through block randomization (1:1). The researchers used a randomization list created on a computer application (https://www.randomizer.org/). Pretest data of the study were collected from patients who consented to participate in the study by two independent researchers who were not involved in the implementation of the study. For assigning each patient to a group, the other team members were called by the same independent researcher, and the subjects were assigned to the groups according to the randomization list created. Two independent researchers conducted the assignment of the participants on the intervention and control groups and the evaluation of the outcome measurement data. Since the researchers conducted the interventions, they were not be blinded. However, the participants were blinded because they did not know the hypotheses of the study and which group they were in.

In the first phase of the study, a web-based education program was developed. For this purpose, the researchers developed a "Web-Based Education Needs Assessment Form for Patients with Cancer" based on a review of the literature. In line with the needs analysis and literature, the research team created a web-based education program. A group of 10 experts evaluated the content of the program, including three oncology physicians, four nursing faculty members, and three nurses.

After obtaining expert opinions, a pilot study was conducted with 10 different patients with cancer who met the sampling criteria. The intelligibility and usability of the program were tested in the pilot study. Patients with cancer included in the first stage of the study were not included in the second stage.

In the second phase of the study, the web-based education program was introduced to the patients with cancer in the intervention group during face-to-face interviews. They were asked to examine the program for at least two hours a week for three months. During the follow-up period, the patients in the intervention group were called twice a week and reminded to use the education program. The researchers get in contact with the patients online via the website. During the follow-up period, the patients contact the research team by calling or writing messages via the website 24/7. An e-mail account was created by the research team using the email system of the university, and it was shared with the patients. The clinical researchers of the team answered the patients' questions via this e-mail account. Within the scope of the study, a new cell phone number was purchased, and the researchers used on a rotating basis to answer patients' questions as a phone response system. During the follow-up, patients' questions were answered on the phone. The control group received routine patient education and routine hospital follow-ups given by Oncology Education Nurses during the three-month follow-up period. In the third month, after the follow-up stage of the study was completed, the post-tests were administered to the patients in the intervention and control groups who came to the hospital for follow-up or treatment. The outcome measures of the study were determined as the symptoms experienced by patients with cancer, quality of life, self-efficacy, and depression levels.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-70 years
* Received at least two cycles of systemic chemotherapy
* Had no verbal communication disorder
* Literate
* Had Internet access
* Use the Internet

Exclusion Criteria:

* Having diagnosed with psychiatric disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Rotterdam Symptom Checklist | 12 week
  The Rotterdam Symptom Checklist is used to evaluate the problems of patients with cancer developing due to the symptoms they experience. The items on the scale are scored between 1 and 4 by using a Likert-type scoring system. The scale consists of 39 items and has 4 sub-dimensions: Physical Symptom Discomfort, Psychological Discomfort, Activity Level, and Quality of Life. The higher the scores obtained from the scale, the greater the distress. Cronbach's alpha value of the scale was determined as 0.88.
EORTC-QLQ-C30 Quality of Life Scale | 12 week
  The EORTC-QLQ-C30 Quality of Life Scale was developed to measure the quality of life of patients with cancer. It includes 30 questions and three sub-dimensions: General Well-Being, Functional Difficulties, and Symptom Control. The maximum score on the scale is 100, and the minimum is 0. High scores on the functional sub-dimension indicate good/healthy functional status, high scores on the symptom sub-dimension indicate high levels of symptoms and/or problems, and high scores on the global health status/quality of life sub-dimension indicate good quality of life.
Strategies Used by Patients to Promote Health | 12 week
  This scale is used to assess the self-confidence of individuals in fulfilling the strategies they use to improve health. It consists of 29 items under 3 sub-dimensions, namely, coping with stress, decision making, and positive behavior development. The scores that can be obtained from the scale range from 29 to 145, and increased scores indicate an increased level of self-efficacy. Cronbach's alpha value of the scale was found as 0.92.
Beck Depression Scale | 12 week
  Beck Depression Scale is a self-assessment scale that measures the symptoms of depression observed in physical, emotional, cognitive, and motivational areas. The purpose of the scale is not to diagnose of depression, but to objectively measure the severity of depressive symptoms. Each of the 21 items on the scale includes four statements numbered 0, 1, 2, and 3. Two of the items on the scale are reserved for emotions, eleven items for cognitions, two items for behavior, five items for somatic symptoms, and one item for interpersonal symptoms. The total score that can be obtained from the scale varies between 0 and 63, and the scores are interpreted as follows: 0-9, no depression; 10-15, mild depression, 16-23 moderate depression, and 24-63 severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Hicran Bektas, PhD, RN, Study Director — Akdeniz University; Hasan S Coskun, Medical Dr, Principal Investigator — Akdeniz University; Fatma Arikan, PhD, RN, Principal Investigator — Akdeniz University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bektas H, Coskun HS, Arikan F, Ozcan K, Tekeli A, Kondak Y, Sezgin MG, Yangec E, Kalav S. Development and evaluation of the efficacy of a web-based education program among cancer patients undergoing treatment with systemic chemotherapy: a randomized controlled trial. Support Care Cancer. 2022 Jul;30(7):6021-6033. doi: 10.1007/s00520-022-07039-w. Epub 2022 Apr 12. PMID 35412076